CLINICAL TRIAL: NCT00174122
Title: Procalcitonin in Diagnosing Bacteremia in the Emergency Department
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361701115
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2006-03-01 (Estimated); Status verified 2004-09

CONDITIONS: Sepsis; Fever
Keywords: Emergency department; Blood culture; Antimicrobial therapy
MeSH Terms: conditions — Sepsis; Fever; Emergencies

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Nowadays, a physician plays a more important role in managing patients with potential infectious complications in the emergency room. Previous studies demonstrated the importance of early and adequate anti-microbial therapy in reducing the mortality and morbidity of patients with severe sepsis. However, in one study, about 6% of clinically significant bacteremic patients were misdiagnosed and discharged from the emergency room. In other studies, about 8.5 to approximately 17% of empirical antibiotic selection was judged inappropriately according to subsequent microbiology, and anti-microbial susceptibility was a result. It reflects the diversity in the presentations of infectious diseases and limited available microbiological reports from the first-line emergency physicians. Timely diagnosis and selection of appropriate antibiotics/treatment in treating those patients challenge an emergency physician more than ever before.

A serum marker, procalcitonin, was recently demonstrated to be a potential indicator in distinguishing between non-infectious and infectious acute inflammatory reactions, viral and bacterial infections, and non-bacteremic and bacteremic infections. It also demonstrates the association with high-mortality risk in patients with severe sepsis. However, some areas remain inconclusive in the clinical application of this potential serum marker.

The investigators designed this prospective study with the following purposes:

1. To clarify the sensitivity and specificity of the serum procalcitonin quantitative test as a clinical indicator of sepsis;
2. To identify the cut-off value of the serum procalcitonin level in sepsis screening among various groups of patients with different co-morbidities;
3. To test the potential role of the procalcitonin quantitative test in identifying occult sepsis in patients with an acute undifferentiated febrile reaction in the emergency room;
4. To test the possibility of the sequential procalcitonin quantitative test as a serological guide of the appropriateness of an empirical antibiotic before the microbiology results are available.

Conclusions in the investigators' study will clarify the clinical application of the serum procalcitonin quantitative test in the differential diagnosis of patients with systemic inflammatory reaction syndrome, the screening of high-risk sepsis patients, and the effectiveness of an empirical antibiotic evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Emergency department patient
* Patient suspected sepsis

Exclusion Criteria:

* Patient less than 15 years of age

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2005-07; Study Completion 2006-06

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Jone Chen, MD, PhD, Study Director — National Taiwan University Hospital
Locations (1):
- Department of Emergency Medicine, National Taiwan University Hospital, Taipei, Taiwan